CLINICAL TRIAL: NCT06938490
Title: A Randomized Multicenter Prospective Study of Colorectal Anastomosis Failures With First Sigmoid or Left Colonic Artery Preservation With D3 Lymphadenectomy (COLAP-D3 - Colorectal Anastomotic Leakage and Arterial Preservation With D3 Lymphadenectomy)
Brief Title: Study of Colorectal Anastomosis Failures With First Sigmoid or Left Colonic Artery Preservation With D3 Lymphadenectomy
Acronym: COLAP-D3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: the BELOOSTROV Clinic of High Technologies (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Beloostrov Clinic High Tech
Record Dates: First submitted 2025-03-26; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer (CRC); Surgery, Colorectal; Oncology
Keywords: Anastomotic leakage; Colorectal cancer (CRC); First sigmoid artery (SA); Left colonic artery (LCA)
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCA preserved (Active Comparator): A group of people with only the left colonic artery preserved
  Interventions: Procedure: Anterior rectal resection with D3-lymphatic dissection
- First SA preserved (Active Comparator): A group of people with only the first sigmoid artery preserved
  Interventions: Procedure: Anterior rectal resection with D3-lymphatic dissection

INTERVENTIONS:
Procedure: Anterior rectal resection with D3-lymphatic dissection — This study aims to determine the incidence of anastomosis failure in the group with first SA and LCA preservation in order to identify the feasibility of manipulation.
  The study is unique in that there is only one study in the world that evaluates the incidence of anastomosis failure with preservation of the first sigmoid and there is no study comparing the groups described in this study.

SUMMARY:
This study is a randomized, controlled trial comparing the short- and long-term outcomes of left colonic artery or first sigmoid artery preservation for rectal surgery. Eligible patients will be randomized to D3-lymphodissection with preservation of the first sigmoid artery or left colonic artery in a 1:1 ratio according to a computer-generated randomization list created in advance (includes removal of 252, 253 l/u groups, 241 groups of distal sigmoid colon sites when the neoplasm is highly located).

The operation involves removal of the tumor with oncologically adequate clearance, adherence to the principles of operation in embryonic layers.

The criterion for performing D3-lymphodissection is visualization of the site of the inferior mesenteric artery (IMA) branching from the aorta. During the surgical intervention, l/u groups 252 and 253 are elevated along the superior rectus artery, the NBA is skeletonized circularly so that there are no l/u and no visible areas of fatty tissue.

In the group with preservation of the left colonic artery, the NBA is isolated, clipped and crossed immediately after the LCA, and in the group with preservation of the first SA, the NBA is skeletonized to the level of the first sigmoid artery, clipped and crossed immediately after the first sigmoid artery . After the intestinal resection stage, a colorectal anastomosis is formed, information on drain placement.

The primary endpoint is to assess the incidence of IA - communication of the intraluminal compartment of the intestine with the extraluminal compartment, anastomosis leakage in the area of the formed anastomosis - which will be performed at 30 days postoperatively and categorized according to the Clavien-Dindo scale. HA can be diagnosed by MRI, CT with proctography, endoscopic examination, or patient examination (if low anastomoses are formed).

Any adverse event in the postoperative period is also classified according to the Clavien-Dindo scale and recorded in the individual patient's chart.

Each patient will have an individual electronic record (eCRF open clinica.), where individual patient data will be entered and where the data obtained will be stored.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. ECOG status is 0-2.
3. Age over 18 years
4. TNM stage according to version VIII T1b-4aN0-2M0 (M1 in case of resectable metastases confirmed by preoperative staging (colonoscopy, chest and abdominal CT).
5. Histologically confirmed adenocarcinoma of the colon, the proximal edge of which is not higher than or equal to 20 cm from the anus
6. Clinical indications for colorectal resection with anastomosis formation

Exclusion Criteria:

1. Medical or psychiatric reasons affecting the patient's decision to participate in the study
2. Pregnancy or breastfeeding
3. Medical conditions contraindicated for surgery
4. Synchronous or metachronous malignancies
5. Acute intestinal obstruction, bleeding or perforation
6. Preplanned obstructive bowel resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 778 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Failure of colorectal anastomoses within 30 days of surgery | 3 years
  The failure of colorectal anastomosis will be registered in the presence of clinical symptoms confirmed by rectal examination (with low anastomoses) and/or MRI

SECONDARY OUTCOMES:
Assessment of radicality of surgery: number of LU removed | 3 years
Long-term results: overall and recurrence-free survival at 1 year, 3 and 5 years, respectively, the percentage of three- and five-year survival in the group where sigmoid artery preservation was performed and where it was clipped. | 3 years
Registration of all deviations from the normal course in the postoperative period | 3 years
Assessment of radicality of surgery: proximal and distal clearance | 3 years
Assessment of radicality of surgery: number of R1 resections | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beloostrov Clinic High Tech, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No